CLINICAL TRIAL: NCT03058874
Title: The Effect of a Dry-weight Probing Guided by Lung Ultrasound on Ambulatory Blood Pressure and Arterial Stiffness in Hemodialysis Patients. A LUST Sub-study.
Brief Title: Effect of Dry-weight Probing Guided by Lung-Ultrasound on Ambulatory Blood Pressure and Arterial Stiffness in Hemodialysis Patients (LUST Sub-Study)
Acronym: LUST ABPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmine Zoccali (Other Government)
Collaborators: Aristotle University Of Thessaloniki (Other); CNR-IBIM Clinical Epidemiology of Renal Diseases and Hypertension Unit, Reggio, Italy (Unknown); University Clinical Centre of Maribor, Slovenia (Unknown)
Responsible Party: Sponsor-Investigator, Carmine Zoccali, MD, FASN, Professor of Nephrology (PG), Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Organization: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELKE 93367
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Hypertension
Keywords: Chronic Kidney Disease; Hemodialysis; Hypertension; Arterial Stifness; Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Renal Dialysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): Standard protocol of fluid management in hemodialysis
  Interventions: Other: Standard protocol of fluid management in hemodialysis
- Active arm (Experimental): Extra-vascular lung water measurements by ultrasound (LW-US)
  Interventions: Device: Extra-vascular lung water measurements by ultrasound

INTERVENTIONS:
Device: Extra-vascular lung water measurements by ultrasound — Lung congestion measured by lung ultrasound (US-B lines) to guide dry-weight probing and UF intensification
  Other Names: Lung Ultrasound Guided Treatment
  Arms: Active arm
Other: Standard protocol of fluid management in hemodialysis — The intervention consists in applying a standard clinical approach for monitoring/tailoring fluid excess in HD patients.
  Arms: Control arm

SUMMARY:
The most common co-morbidity accompanying Chronic Kidney Disease (CKD) is hypertension, which appears in approximately 80% of all patients with renal dysfunction, whereas its prevalence in general population is remarkably lower appearing in approximately 30% of adults.Defining hypertension in ESRD patients under maintenance dialysis is a challenging procedure. Ambulatory blood pressure monitoring (ABPM) is considered the "gold standard" for the diagnosis of hypertension in hemodialysis patients over the last years. The major pathophysiologic mechanism underlying hypertension development in patients with ESRD under hemodialysis is water and sodium overload.

Identifying an accurate and objective method of dry weight evaluation has been a matter of intensive nephrology research for more than two decades. Assessment of the water balance in hemodialysis patients on the basis of common clinical criteria (e.g. leg or face swelling or signs of lung congestion) is a subjective method with limited reliability, despite its widespread use. Recently, a novel technique has been developed to quantify water excess by conducting an ultrasound lung scan. Pilot studies have shown significant changes in lung water in hemodialysis patients according to body weight changes during interdialytic days and dialysis sessions. Moreover, results from previous studies indicate significant benefits from dry weight probing with regards to blood pressure (BP).

The clinical application of a lung-ultrasound-based volume control strategy in hemodialysis patients is currently being tested by the randomized study entitled "Lung water by ultrasound guided treatment to prevent death and cardiovascular complications in high risk end stage renal disease patients with cardiomyopathy (The LUST Study)". This clinical trial aims at evaluating whether the use of the number of US-B lines could be used as a biomarker to guide a per-protocol intensification of ultrafiltration (UF) in order to reduce volume overload, improve cardiac function and prolong survival.

Cardiovascular disease in patients with CKD is attributed to a spectrum of structural and functional alterations of the large and the small branches of the arterial tree. The most important process in patients with advanced CKD is that of arteriosclerosis, which is developed in parallel to atherosclerosis and is typically associated with impaired cushioning function of the aorta and the large conduit arteries. Accelerated arterial stiffening is involved in the development of isolated systolic hypertension, left ventricular hypertrophy (LVH) and congestive heart failure (CHF), which predispose to arrhythmias and sudden cardiac death. In the context of the phenomenon of "aortic-to-brachial BP amplification", systolic BP (SBP) and pulse pressure (PP) conventionally measured at the level of brachial artery are higher than the relevant pressures in the ascending aorta. Due to extreme elevation of arterial stiffness, BP amplification is disturbed in patients with ESRD. Prospective cohort studies have demonstrated that elevated central PP, wave reflections and arterial stiffness, as well as, reduced PP amplification represent strong and independent predictors of all-cause and cardiovascular mortality in hemodialysis patients. On this basis, estimation of central BP indices appears as an important tool towards optimisation of cardiovascular risk stratification in ESRD as well as in other diseased populations.

Until recently, available devices for ABPM evaluated BP levels only at the level of brachial artery. The newly developed Mobil-O-Graph NG (IEM, Stolberg, Germany) provides the ability to monitor central aortic pressure and indices of vascular resistance, such as wave reflections (augmentation index, AIx) and arterial stiffness (pulse wave velocity, PWV).This device has recently been validated in hemodialysis patients and showed comparable performance with the widely used tonometric SphygmoCor device (ArtCor, Sydney, Australia). Accumulated evidence over central BP and PWV in hemodialysis patients derives mostly from studies that included only static pre-dialysis and post-dialysis measurements. However, variations of BP levels during intra- and interdialytic intervals combined with the superiority of aortic BP measurements, as analysed above, indicate that ambulatory monitoring of central BP is the best available method.

This study aims for the first time to evaluate the outcome of a treatment strategy for dry weight probing, based on volume overload quantification with lung ultrasound, on 48-hour peripheral systolic BP, aortic BP and arterial stiffness in hemodialysis hypertensive patients.

This is a Lust Sub-Study. Additional information can be found at: NCT02310061.

DETAILED DESCRIPTION:
Patient selection and study preparations

Potentially eligible hemodialysis patients, not fitting the exclusion criteria, will provide written informed consent and will be evaluated for the diagnosis of hypertension. If patients are treated with antihypertensive therapy, a brief-wash out from medications period will take place and home BP will be monitored up to a maximum of 4 weeks. During this period BP ≥160/110 mmHg will be a threshold for further medication withdrawal.

Hypertension diagnosis will be based on mean BP values ≥135/85 mmHg with home BP monitoring the days after the mid and last dialysis of the week for 2 consecutive weeks using a validated self-inflating automatic oscillometric device (cuff with bladder size encircling at least 80% of arm circumference and covering two thirds of arm length). Every patient will be asked to conduct both morning and evening BP measurements at the level of brachial artery after 5 min of rest and with two measurements per occasion taken 2 min apart according to the European Society of Hypertension 2013 guidelines. The mean of the last measurements would be used.

Study period

A total number of 70 eligible patients undergoing hemodialysis in the Hemodialysis Unit of the Department of Nephrology, Hippokration Hospital, Aristotle University of Thessaloniki, Greece and in affiliated Hemodialysis Units in Northern Greece, as well in the Hemodialysis Units of the Department of Nephrology University Clinical Centre Maribor, Slovenia will participate in the study. In all potentially eligible patients full medical history, as well as demographic characteristics and drug treatment will be recorded, followed by a detailed physical examination. Patients that meet the inclusion and exclusion criteria, will be randomized with a ratio of 1:1 into two equal groups consisting of 35 patients. In the intervention group a specific treatment strategy for dry-weight reduction will be applied guided by lung ultrasound, whereas in the control group standard-of-care treatment will be applied guided by conventional clinical criteria. Blood samples for hematological and biochemical laboratory tests will be collected at baseline prior to a mid-week dialysis session; these tests will correspond to the routine monthly laboratory tests of the patients.

In the intervention group UF regimen and dry-weight will be guided by the number of pre-dialysis US-B lines measured by lung ultrasound prior to a mid-week dialysis session. In patients who will be included in both the main study (LUST) and the present sub-study (i.e. additional inclusion criteria of LUST study: history of myocardial infarction with or without ST elevation or unstable angina, acute coronary syndrome documented by ECG recordings and cardiac troponins or stable angina pectoris with documented coronary artery disease by prior coronary angiography or ECG or dyspnea class III-IV NYHA), a total number of ≥15 US-B lines indicates moderate to severe lung congestion; UF will be intensified in these patients. They will undergo dry-weight reduction less than 0.2 kg/session (0.6 kg/week) with a maximum UF rate ≤10 ml/kg/h, so that episodes of hemodynamic instability and hypotension are minimized. If needed longer and/or additional dialysis sessions will be applied to a maximum of 5 hours/session or 4 sessions/week. US-B lines measurements will be repeated at least once a week (before and after a mid-week dialysis session) until the treatment goal is achieved (<15 US-B lines) over a period of 8 weeks. Thereafter, lung ultrasound will be conducted once a month. In patients without pulmonary congestion at pre-dialysis baseline (<15 US-B lines), no UF intensification will be applied and US-B lines will be measured on a weekly basis. Patients in the intervention group with <15 US-B lines at baseline who will develop clinical signs of pulmonary congestion and/or ≥15 US-B lines at any time will be treated according to those with lung congestion at baseline. In patients who will be included only in the present sub-study, and are expected to have hypertension with better cardiac function and, possibly, less degree of lung congestion compared to the typical subjects of the main LUST study, UF will be intensified on the basis of a total number of ≥5 US-B lines which indicates mild to moderate lung congestion. These patients will also undergo careful dry-weight reduction less than 0.2 kg/session (0.6 kg/week) with a maximum UF rate ≤10 ml/kg/h, so that episodes of hemodynamic instability and hypotension are minimized. If needed longer and/or additional dialysis sessions will be applied to a maximum of 5 hours/session or 4 sessions/week. US-B lines measurements will be repeated at least once a week (before and after a mid-week dialysis session) until the treatment goal is achieved (<5 US-B lines) over a period of 8 weeks. Thereafter, lung ultrasound will be conducted once a month. In patients without pulmonary congestion at pre-dialysis baseline (<5 US-B lines), no UF intensification will be applied and US-B lines will be measured on a weekly basis. Patients in the intervention group with <5 US-B lines at baseline who will develop clinical signs of pulmonary congestion and/or ≥5 US-B lines at any time will be treated according to those with lung congestion at baseline.

Reduction of post-dialysis weight with UF intensification to achieve treatment goal will be pursued for 8 weeks. During this period BP should be maintained in levels <160/110 mmHg. If BP exceeds these levels, per protocol drug therapy will be initiated. As a first step, carvedilol per os will be administered on a starting dose of 3.125 mg b.i.d. up to a maximum tolerated dose (≤25 mg b.i.d.) until BP levels are <160/110 mmHg or until patient experiences signs of bradycardia (HR <60 bpm) or other adverse effects. As a second step of drug therapy, irbesartan will be initiated on a starting dose of 75 mg daily up to maximum tolerated dose (≤300 mg daily) until BP levels are <160/110 mmHg or any adverse effects are presented. Finally, amlodipine on a starting dose of 5 mg daily up to maximum tolerated dose (≤10 mg daily) will be administered on failure of the two previous steps to achieve BP levels <160/110 mmHg. If BP is still not controlled at goal, any antihypertensive class can be added according to treating physician's choice.

In the control group follow-up, dry-weight and UF regimen will be guided only by conventional clinical and laboratory criteria. Blood pressure and blood pressure changes over time, pedal edema, presence or absence of dyspnea, body weight gain between dialysis and hemodynamic instability during dialysis session will be some of the clinical criteria that will determine possible post-dialysis weight adjustments in these patients. The use of lung ultrasound to estimate lung congestion will not be allowed in these patients. A threshold of BP 160/110 mmHg will be set for the first 8 weeks of the study. If BP exceeds these levels, per protocol drug therapy will be initiated as mentioned in the intervention group.

After 8 weeks of treatment, per protocol drug therapy will be performed in patients from both study groups, aiming at maintaining Home BP levels <135/85 mmHg.

The primary and secondary measurements of the study will be carried in prespecified time-points that are listed below:

Study-Point 1:

Participants in the study will be asked to come to their dialysis unit 30 min before the start of the first or second dialysis of the week. A Mobil-O-Graph monitor with a cuff of appropriate size will be fitted to and BP will be recorded for 48 hours. The device will be programmed to collect data every 20 minutes, except for 23:00 to 07:00 (data collection every 30 minutes). An ABPM would be considered successful if >80% of recordings are valid with no more than two non-consecutive day hours (07.00-23.00 hours) with fewer than two valid measurements, and no more than one night hour (23.00-07.00 hours without valid recording, according to standard recommendations for ABPM. Patients with unsuccessful 24-hour ABPM will repeat the measurement a week later.

Participants in the study will further come to the echocardiography unit on the first or the second interdialytic day of the week (Tuesday or Thursday for patients on M-W-F schedule and Wednesday or Friday for patients on T-T-S schedule) exactly 24 hours after the scheduled starting time of the previous dialysis session. All study participants will undergo an echocardiography study, as well as US-B lines measurement with lung ultrasound. Body composition would be estimated with the use of Bioelectrical Impedance Analysis. PWV and AIx recordings with the Sphygmocor device would be taken. The results from this echocardiographic study and 48-hour ABPM will be used as the baseline reference..

Following echocardiographic assessment, patients will be randomized in 1:1 ratio in the intervention and control arms with permuted blocks of 4 subjects, using a computer-generated randomization schedule stratified by sex and center.

Participants in the study will be asked to come to their dialysis unit one hour earlier than their second (Wednesday or Thursday) or the third (Friday or Saturday) dialysis session of the week is scheduled, following at least a 8-hour fast and without having received their morning medication. The ABPM device will be removed and checked for completeness. Patients with unsuccessful 48-hour ABPM will repeat the measurement and all further evaluations a week later. Body weight will be measured with the use of validated electronic weighting scales. Height will be also evaluated for the BMI calculation. Office blood pressure measurements will be acquired after 5 min of rest (sitting posture) with the use of a validated oscillometric device or standard mercury sphygmomanometer at the level of brachial artery in the contralateral arm of the side where vascular access is located. Venous blood specimens will be collected for routine hematological and biochemical laboratory testing, as mentioned before. A lung ultrasound will be conducted in all study participants in the intervention group using the GE VScan lung ultrasound device, 15 minutes before hemodialysis session initiation. With patient in a lying posture pre-dialysis US-B lines will be measured in both lungs, while the transducer is placed vertically from the second up to the fifth intercostal space consecutively, along the parasternal, the mid-clavear, the anterior axillary and the mid axillary lines. All measurements will be performed in a quiet room with controlled air temperature (approximately 22 ° C) The sum of the US-B lines produces a score (US-B lines score) and UF regimen will be guided accordingly. In patients who will be include in both the main LUST study and the present sub-study with ≥15 US-B lines and in patients who will be included only in this sub-study with ≥5 US-B lines, UF will be intensified and dry-weight will be reduced according to the value of US-B lines score over a period of 8 weeks (Figure 2). Thresholds in dry-weight reduction and UF rates will be applied and if needed longer and/or additional dialysis sessions will be conducted as mentioned before. In the control arm standard-of-care treatment will be applied guided by conventional clinical criteria.

Afterwards all study participants from both arms will undergo their scheduled dialysis session.

Over the period of the first 8 weeks of the study US-B lines measurements with lung ultrasound will be repeated at least once a week (before and after a mid-week dialysis session) in all patients in the active arm. During this period per protocol drug therapy will be initiated if BP exceeds a threshold of home BP 160/110 mmHg.

Study Point 2:

Two months (8 weeks) after baseline all patients will be subjected again in the examinations described at Study Point 1 (i.e. 48-hour ABPM, echocardiography, bioimpedance analysis and pulse wave tonometry) exactly in the same manner with regards to the scheduled hemodialysis sessions.

If treatment goal is achieved during this post-dialysis US-B lines measurement, lung ultrasounds will be conducted once a month from this point on. Patients in the intervention group who have achieved the treatment goal of post-dialysis US-B lines score at previous evaluations and who will develop clinical signs of pulmonary congestion and/or ≥15 or ≥5 US-B lines according to the patients' stratification at any time will be treated according to those with lung congestion at baseline. A threshold of Home BP <135/85 mmHg will be set after this point and when needed the same per protocol drug therapy will be performed in patients from both study groups.

Study Point 3:

One year after their first evaluation all patients will undergo all examinations described in baseline, with a similar order.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Dialysis vintage > 3 months
* A history of hypertension, confirmed by valid Home BP readings
* Written consent to take part in the study

Exclusion Criteria:

* Cancer or other advanced non cardiac disease or co-morbidity (e.g. end-stage liver failure) imposing a very poor short-term prognosis
* Active infections or relevant inter-current disease
* Inadequate lung scanning and echocardiographic studies
* Hemodynamic instability during dialysis session that require intravenous fluid administration to restore BP, in over 30% of sessions during the past 3 months
* Patients with modification of their dry weight and antihypertensive treatment during one month prior to study enrolment
* Nonfunctional arteriovenous fistula in the contralateral arm of the one used as vascular access for the hemodialysis session
* Patients with Home BP readings >180/110 mmHg
* Patients with history of drug or alcohol abuse or known severe mental disorder
* Pregnancy at study entry or during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Difference between groups in changes in 48-hour Brachial Systolic Blood Pressure, obtained with the Mobilograph device | 0, 2, 12 months

SECONDARY OUTCOMES:
Difference between groups in changes in 48-hour Brachial Diastolic Blood Pressure, obtained with the Mobilograph device | 0, 2, 12 months
Difference between groups in changes in 48-hour Aortic Systolic Blood Pressure, obtained with the Mobilograph device | 0, 2, 12 months
Difference between groups in changes in 48-hour Aortic Diastolic Blood Pressure, obtained with the Mobilograph device | 0, 2, 12 months
Difference between groups in changes in ambulatory pulse pressure (PP), obtained with the Mobilograph device | 0, 2, 12 months
Difference between groups in changes in ambulatory augmentation index (AIx), obtained with the Mobilograph device | 0, 2, 12 months
Difference between groups in changes in ambulatory pulse wave velocity (PWV), obtained with the Mobilograph device | 0, 2, 12 months
Difference between groups in changes in echocardiographic indices of left ventricular function | 0, 2, 12 months
Difference between groups in changes in Body composition assessed with bioelectrical impedance analysis | 0, 2, 12 months
Difference between groups in changes in PWV, obtained with the Sphygmocor device | 0, 2, 12 months
Difference between groups in changes in AIx, obtained with the Sphygmocor device | 0, 2, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pantelis A Sarafidis, MD, MSc, PhD, Principal Investigator — Department of Nephrology, Hippokration Hospital, Aristotle University of Thessaloniki
Locations (2):
- Aristotle University, Thessaloniki, Greece
- University Clinical Centre of Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coresh J, Byrd-Holt D, Astor BC, Briggs JP, Eggers PW, Lacher DA, Hostetter TH. Chronic kidney disease awareness, prevalence, and trends among U.S. adults, 1999 to 2000. J Am Soc Nephrol. 2005 Jan;16(1):180-8. doi: 10.1681/ASN.2004070539. Epub 2004 Nov 24. PMID 15563563
- [Background] Sarafidis PA, Li S, Chen SC, Collins AJ, Brown WW, Klag MJ, Bakris GL. Hypertension awareness, treatment, and control in chronic kidney disease. Am J Med. 2008 Apr;121(4):332-40. doi: 10.1016/j.amjmed.2007.11.025. PMID 18374693
- [Background] Georgianos PI, Sarafidis PA, Zoccali C. Intradialysis Hypertension in End-Stage Renal Disease Patients: Clinical Epidemiology, Pathogenesis, and Treatment. Hypertension. 2015 Sep;66(3):456-63. doi: 10.1161/HYPERTENSIONAHA.115.05858. Epub 2015 Jul 6. No abstract available. PMID 26150436
- [Background] Agarwal R. Volume-associated ambulatory blood pressure patterns in hemodialysis patients. Hypertension. 2009 Aug;54(2):241-7. doi: 10.1161/HYPERTENSIONAHA.109.136366. Epub 2009 Jun 15. PMID 19528362
- [Background] Agarwal R, Alborzi P, Satyan S, Light RP. Dry-weight reduction in hypertensive hemodialysis patients (DRIP): a randomized, controlled trial. Hypertension. 2009 Mar;53(3):500-7. doi: 10.1161/HYPERTENSIONAHA.108.125674. Epub 2009 Jan 19. PMID 19153263
- [Background] Zoccali C, Tripepi R, Torino C, Tripepi G, Mallamaci F. Moderator's view: Ambulatory blood pressure monitoring and home blood pressure for the prognosis, diagnosis and treatment of hypertension in dialysis patients. Nephrol Dial Transplant. 2015 Sep;30(9):1443-8. doi: 10.1093/ndt/gfv241. Epub 2015 May 28. PMID 26022727
- [Background] Sarafidis PA, Georgianos PI, Karpetas A, Bikos A, Korelidou L, Tersi M, Divanis D, Tzanis G, Mavromatidis K, Liakopoulos V, Zebekakis PE, Lasaridis A, Protogerou AD. Evaluation of a novel brachial cuff-based oscillometric method for estimating central systolic pressure in hemodialysis patients. Am J Nephrol. 2014;40(3):242-50. doi: 10.1159/000367791. Epub 2014 Oct 11. PMID 25322847
- [Background] London GM, Cohn JN. Prognostic application of arterial stiffness: task forces. Am J Hypertens. 2002 Aug;15(8):754-8. doi: 10.1016/s0895-7061(02)02966-7. PMID 12160201
- [Background] London GM, Pannier B. Arterial functions: how to interpret the complex physiology. Nephrol Dial Transplant. 2010 Dec;25(12):3815-23. doi: 10.1093/ndt/gfq614. Epub 2010 Oct 14. PMID 20947536
- [Background] Karpetas A, Sarafidis PA, Georgianos PI, Protogerou A, Vakianis P, Koutroumpas G, Raptis V, Stamatiadis DN, Syrganis C, Liakopoulos V, Efstratiadis G, Lasaridis AN. Ambulatory recording of wave reflections and arterial stiffness during intra- and interdialytic periods in patients treated with dialysis. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):630-8. doi: 10.2215/CJN.08180814. Epub 2015 Jan 29. PMID 25635033
- [Background] Zoccali C, Mallamaci F. Arterial Stiffness as a Cardiovascular Risk Factor in Stage 5D Chronic Kidney Disease Patients: An Age Affair. Am J Nephrol. 2017;45(1):69-71. doi: 10.1159/000453339. Epub 2016 Nov 30. No abstract available. PMID 27898424
- [Background] Mallamaci F, Benedetto FA, Tripepi R, Rastelli S, Castellino P, Tripepi G, Picano E, Zoccali C. Detection of pulmonary congestion by chest ultrasound in dialysis patients. JACC Cardiovasc Imaging. 2010 Jun;3(6):586-94. doi: 10.1016/j.jcmg.2010.02.005. PMID 20541714
- [Background] Torino C, Gargani L, Sicari R, Letachowicz K, Ekart R, Fliser D, Covic A, Siamopoulos K, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Gueler F, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Siriopol D, Balafa O, Shavit L, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. The Agreement between Auscultation and Lung Ultrasound in Hemodialysis Patients: The LUST Study. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):2005-2011. doi: 10.2215/CJN.03890416. Epub 2016 Sep 22. PMID 27660305
- [Background] Gargani L, Sicari R, Raciti M, Serasini L, Passera M, Torino C, Letachowicz K, Ekart R, Fliser D, Covic A, Balafa O, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Shavit L, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Kraemer TD, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Onofriescu M, Zarzoulas F, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. Efficacy of a remote web-based lung ultrasound training for nephrologists and cardiologists: a LUST trial sub-project. Nephrol Dial Transplant. 2016 Dec;31(12):1982-1988. doi: 10.1093/ndt/gfw329. Epub 2016 Sep 26. PMID 27672089
- [Derived] Loutradis C, Papadopoulos CE, Sachpekidis V, Ekart R, Krunic B, Karpetas A, Bikos A, Tsouchnikas I, Mitsopoulos E, Papagianni A, Zoccali C, Sarafidis P. Lung Ultrasound-Guided Dry Weight Assessment and Echocardiographic Measures in Hypertensive Hemodialysis Patients: A Randomized Controlled Study. Am J Kidney Dis. 2020 Jan;75(1):11-20. doi: 10.1053/j.ajkd.2019.07.025. Epub 2019 Nov 12. PMID 31732234
- See also: The LUST Study (NCT02310061) — https://clinicaltrials.gov/ct2/show/study/NCT02310061?show_desc=Y